CLINICAL TRIAL: NCT00854932
Title: Effect of Procalcitonin-guided Decision Making on Duration of Antibiotic Therapy in Suspected Neonatal Early-onset Sepsis: Multicenter Prospective Randomized Intervention Study
Brief Title: Neonatal Procalcitonin Intervention Study
Acronym: NeoPInS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Kantonsspital Winterthur KSW (Other); Triemli Hospital (Other); Kantonsspital Graubuenden (Other); Insel Gruppe AG, University Hospital Bern (Other); Jeroen Bosch Ziekenhuis, s'-Hertogenbosch (Unknown); Amsterdam UMC, location VUmc (Other); Reinier de Graaf Groep (Other); Erasmus Medical Center (Other); Thomayer University Hospital (Other); Flevo Ziekenhuis, Almere (Unknown); Atrium Medisch Centrum, Heerlen (Unknown); Ijssalland Ziekenhuis, Capelle aan den Ijssel (Unknown); Sint Franciscus Gasthuis (Other); Vlietland Ziekenhuis (Other); McMaster University (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Stocker Martin, MD, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoPInS
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Sepsis
Keywords: procalcitonin; sepsis; newborn; intervention study
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCT group (Experimental): In the PCT group, if infection is considered to be unlikely or possible, antibiotic therapy is discontinued when two consecutive PCT values are within the normal range.Antibiotic therapy can be continued despite fulfilled criteria at the discretion of the attending physician. These divesions from the stopping rules will be reported for further analysis.
  Interventions: Other: Procalcitonin-guided decision making
- Standard group (No Intervention): The duration of antibiotic treatment in the standard group is based on the attending physician's assessment of the risk of classification: infection unlikely for 36-72 hours, infection possible for 5-7 days, infection probable of proven for 7-21 days depending on clinical course, laboratory values and positive cultures.

INTERVENTIONS:
Other: Procalcitonin-guided decision making — In the PCT group, if infection is considered to be unlikely or possible, antibiotic therapy is discontinued when two consecutive PDT values are within the normal range.
  Other Names: Procalcitonin-guided duration of antibiotic therapy
  Arms: PCT group

SUMMARY:
In neonates, clinical signs and symptoms associated with early-onset sepsis are non-specific and currently available tests have poor positive and negative predictive values. The investigators hypothesize that procalcitonin (PCT) has a reliable negative predictive values to allow a reduction in duration of empiric antibiotic therapy in suspected neonatal early-onset sepsis with unchanged outcome. This study is designed as a multi-center, prospective, randomized intervention trial. The duration of antibiotic therapy in the standard group is based on the attending physician's assessment of the probability of infection during hospitalisation. In the PCT group, if infection is considered to be unlikely or possible, antibiotic therapy is discontinued when two consecutive PCT values are within the normal range.

DETAILED DESCRIPTION:
Detailed description according our pilot study (see reference). This trial is designed to exclude a difference in rate of re-infection or death greater than 2%. Assuming a 2% reinfection/death rate in each group, 770 patients are required for a power of 80% at alpha=0.05. To allow for some unevaluable cases 800 per group will be included. Based on the data of the pilot study (see reference), with a number of 770 per group a difference between mean antibiotic therapy durations of 10 hours can be detected at two-sided alpha of 0.05 with a power of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Term and near term infants with a gestational age > 34 weeks
* Suspected sepsis in the first 3 days of life requiring empiric antibiotic therapy
* Parental consent

Exclusion Criteria:

* Surgery in the first week of life
* Severe congenital malformations

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1600 (Estimated)
Dates: Start 2009-06; Primary Completion 2015-05 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The absolute reduction of the duration of antibiotic therapy with unchanged outcome | 1 month
  Unchanged outcome = proportion of infants with a recurrence of infection requiering additional courses of antibiotic therapy within 72 hours after ending antibiotic therapy and/or death in the first month of life

SECONDARY OUTCOMES:
Duration of hospitalisation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stocker, MD, Principal Investigator — Kantonsspital Luzern, Switzerland
Locations (1):
- children's Hospital of Lucerne, Lucerne, Switzerland

REFERENCES:
- [Background] Stocker M, Fontana M, El Helou S, Wegscheider K, Berger TM. Use of procalcitonin-guided decision-making to shorten antibiotic therapy in suspected neonatal early-onset sepsis: prospective randomized intervention trial. Neonatology. 2010;97(2):165-74. doi: 10.1159/000241296. Epub 2009 Sep 24. PMID 19776651
- [Background] Stocker M, Hop WC, van Rossum AM. Neonatal Procalcitonin Intervention Study (NeoPInS): Effect of Procalcitonin-guided decision making on duration of antibiotic therapy in suspected neonatal early-onset sepsis: A multi-centre randomized superiority and non-inferiority Intervention Study. BMC Pediatr. 2010 Dec 8;10:89. doi: 10.1186/1471-2431-10-89. PMID 21143869
- [Derived] Stocker M, Daunhawer I, van Herk W, El Helou S, Dutta S, Schuerman FABA, van den Tooren-de Groot RK, Wieringa JW, Janota J, van der Meer-Kappelle LH, Moonen R, Sie SD, de Vries E, Donker AE, Zimmerman U, Schlapbach LJ, de Mol AC, Hoffmann-Haringsma A, Roy M, Tomaske M, Kornelisse RF, van Gijsel J, Plotz FB, Wellmann S, Achten NB, Lehnick D, van Rossum AMC, Vogt JE. Machine Learning Used to Compare the Diagnostic Accuracy of Risk Factors, Clinical Signs and Biomarkers and to Develop a New Prediction Model for Neonatal Early-onset Sepsis. Pediatr Infect Dis J. 2022 Mar 1;41(3):248-254. doi: 10.1097/INF.0000000000003344. PMID 34508027
- [Derived] Stocker M, van Herk W, El Helou S, Dutta S, Fontana MS, Schuerman FABA, van den Tooren-de Groot RK, Wieringa JW, Janota J, van der Meer-Kappelle LH, Moonen R, Sie SD, de Vries E, Donker AE, Zimmerman U, Schlapbach LJ, de Mol AC, Hoffman-Haringsma A, Roy M, Tomaske M, Kornelisse RF, van Gijsel J, Visser EG, Willemsen SP, van Rossum AMC; NeoPInS Study Group. Procalcitonin-guided decision making for duration of antibiotic therapy in neonates with suspected early-onset sepsis: a multicentre, randomised controlled trial (NeoPIns). Lancet. 2017 Aug 26;390(10097):871-881. doi: 10.1016/S0140-6736(17)31444-7. Epub 2017 Jul 12. PMID 28711318